CLINICAL TRIAL: NCT06908122
Title: Validity of Laboratory Biomarkers in Diagnosis of Nonalcoholic Fatty Liver Disease (NAFLD) and It's Consequences
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahy nour Zoghby Abd elhi, assisstant lecturer, Assiut University
Other Study IDs: FAM.AssiutU
Record Dates: First submitted 2025-03-11; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: laboratory biomarkers in the diagnosis of NAFLD disease — All included patients will be assessed as follows:
  1. Questionnaire: different questionnaire variables extrapolated from study published by Xin Li, 2024, Bao et al., 2024 (8), (9).The questionnaire will be divided into six parts: First section includes demographic characteristics of patients as (name , age, gender, occupation, educational level and special habits) The second section includes chronic diseases-related questions and drug administration as if a patient were diagnosed with chronic disease, on treatment and drugs used.
  The third section for assessment of dietary lifestyle includes:
  nutrition adherence to Mediterranean will be assessed by a validated 17-item MedDiet adherence questionnaire, which all participants will answer. A score will be given for each met objective: 1 (compliance) or 0 (non-compliance).
  The counseling session will be about the Mediterranean diet program, and a brochure will be given to each patient.

SUMMARY:
The validity of laboratory biomarkers in the diagnosis of NAFLD is still not established, and adherence to a healthy dietary lifestyle for those patients in our community is not well studied.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is characterized by excessive hepatic fat accumulation, associated with insulin resistance, and defined as the histological presence of steatosis in >5% hepatocytes.

NAFLD is an umbrella terminology incorporating a spectrum of liver diseases ranging from simple steatosis (nonalcoholic fatty liver), steatohepatitis (nonalcoholic steatohepatitis, NASH), and cirrhosis. NAFLD is also the leading cause of liver cirrhosis, hepatocellular carcinoma, and death.

Early diagnosis and assessment of NAFLD and liver fibrosis are essential for monitoring disease progression and selecting the best treatment options for affected individuals.

Given that liver biopsy had considerable disadvantages, there was a dire need for genuine noninvasive methods for NAFLD detection and risk assessment. The serum markers and other indicators is valuable for screening diseases due to their convenience, low cost, and accuracy of diagnosis Unhealthy dietary composition is an important factor in the progression of non- alcoholic fatty liver disease. Many studies surround the benefits of a Mediterranean diet in conditions such as metabolic syndrome, T2DM, and cardiovascular disease; such conditions often coexist and have a pathophysiological link with NAFLD.

The Mediterranean diet (MeD) is defined as a plant-based diet characterized by a high intake of fruits and vegetables, legumes, whole grains, and a high ratio of monounsaturated fatty acids (MUFA), which is associated with a lower risk of many chronic diseases

ELIGIBILITY:
Inclusion Criteria:

* All adult patients attending outpatient clinics characterized by an age over 18 years.
* Patients diagnosed as NAFLD.

Exclusion Criteria:

* Patients younger than 18 years old.
* Patients diagnosed with viral hepatitis to avoid other causes of liver fibrosis. .
* Patients with alcoholic fatty liver (more than three standard drinks per day for men or more than two standard drinks per day for women).
* Patients receiving treatment with drugs known to promote liver steatosis (for example, tamoxifen, amiodarone, estrogen, or corticosteroids).
* Patients with malignant tumors or other severe organ dysfunction diseases.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients diagnosed as having NAFLD attend outpatient clinics characterized by an age over 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Validity of lab biomarkers in the diagnosis of nonalcoholic fatty liver disease (NAFLD) and it's consequences in comparison with abdominal ultrasound and fibroscan. | 1 year
  different laboratory ratio will be calculated to assess validity of different laboratory markers in diagnosis of NAFLD

SECONDARY OUTCOMES:
dietary life style and conduct of Mediterranean diet programme counseling for NAFLD patients attending Assiut university hospitals | one year
  -nutrition adherence to Mediterranean will be assessed by a validated 17-item MedDiet adherence questionnaire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ko E, Yoon EL, Jun DW. Risk factors in nonalcoholic fatty liver disease. Clin Mol Hepatol. 2023 Feb;29(Suppl):S79-S85. doi: 10.3350/cmh.2022.0398. Epub 2022 Dec 14. PMID 36517003
- [Background] Han SK, Baik SK, Kim MY. Non-alcoholic fatty liver disease: Definition and subtypes. Clin Mol Hepatol. 2023 Feb;29(suppl):S5-S16. doi: 10.3350/cmh.2022.0424. Epub 2022 Dec 28. PMID 36577427
- [Background] Montemayor S, Mascaro CM, Ugarriza L, Casares M, Llompart I, Abete I, Zulet MA, Martinez JA, Tur JA, Bouzas C. Adherence to Mediterranean Diet and NAFLD in Patients with Metabolic Syndrome: The FLIPAN Study. Nutrients. 2022 Aug 3;14(15):3186. doi: 10.3390/nu14153186. PMID 35956364
- [Background] George ES, Reddy A, Nicoll AJ, Ryan MC, Itsiopoulos C, Abbott G, Johnson NA, Sood S, Roberts SK, Tierney AC. Impact of a Mediterranean diet on hepatic and metabolic outcomes in non-alcoholic fatty liver disease: The MEDINA randomised controlled trial. Liver Int. 2022 Jun;42(6):1308-1322. doi: 10.1111/liv.15264. Epub 2022 Apr 26. PMID 35357066
- [Background] Doustmohammadian A, Clark CCT, Maadi M, Motamed N, Sobhrakhshankhah E, Ajdarkosh H, Mansourian MR, Esfandyari S, Hanjani NA, Nikkhoo M, Zamani F. Favorable association between Mediterranean diet (MeD) and DASH with NAFLD among Iranian adults of the Amol Cohort Study (AmolCS). Sci Rep. 2022 Feb 8;12(1):2131. doi: 10.1038/s41598-022-06035-8. PMID 35136128